CLINICAL TRIAL: NCT01715311
Title: A Randomized, Double-blind Placebo-controlled Study to Compare the Efficacy of Indacaterol With That of Placebo in Patients With COPD Who Have Not Previously Received Maintenance COPD Medication, Using Blinded Tiotropium as Active Control
Brief Title: Comparison of Indacaterol With That of Placebo in 'Maintenance naïve' Patients With COPD Using Blinded Tiotropium as Active Control
Acronym: INITIATE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: withdrawn prior to patient recruitment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2425; 2012-001536-59 (EudraCT Number)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2013-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Chronic obstructive pulmonary disease; indacaterol; tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Tiotropium Bromide; Dry Powder Inhalers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Indacaterol (Experimental): Indacaterol once daily
  Interventions: Drug: Indacaterol; Drug: Placebo to indacaterol
- Placebo (Placebo Comparator): Placebo for indacaterol and placebo for tiotropium once daily
  Interventions: Drug: Placebo to tiotropium; Drug: Placebo to indacaterol
- Tiotropium (Active Comparator): Tiotropium
  Interventions: Drug: Placebo to tiotropium; Drug: Tiotropium

INTERVENTIONS:
Drug: Indacaterol — Indacaterol once daily via single-dose dry powder inhaler
  Arms: Indacaterol
Drug: Placebo to tiotropium — Placebo to tiotropium capsules for inhalation once daily
  Arms: Placebo; Tiotropium
Drug: Tiotropium — Tiotropium capsules for inhalation once daily
  Other Names: Tiotropium 18 mcg od via single-dose dry powder inhaler
  Arms: Tiotropium
Drug: Placebo to indacaterol — Placebo to indacaterol capsules for inhalation once daily
  Arms: Indacaterol; Placebo

SUMMARY:
This study will compare the efficacy of indacaterol versus placebo (i.e., rescue medication only) and tiotropium in patients with Chronic Obstructive Pulmonary Disease (COPD) who have not received maintenance COPD medication for at least 12 months prior to entry (described hereafter as "maintenance naïve", see inclusion criteria).

DETAILED DESCRIPTION:
The purpose is to provide efficacy data comparing the long-acting beta-2 agonist, indacaterol, with short-acting rescue therapy in maintenance-naive patients belonging to GOLD 2011 Groups A and B.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable Chronic Obstructive Pulmonary Disease (COPD) Groups A or B according to GOLD 2011.
* Patients with a post-bronchodilator Forced Expiratory Volume in one second (FEV1) ≥50% and <80% of the predicted normal, and post-bronchodilator FEV1/ Forced Vital Capacity (FVC) < 0.7
* Patients with no record of receipt of maintenance medication for COPD.
* Patients with a mMRC dyspnea score ≥1 at Visit 2.
* Current or ex-smokers who have a smoking history of at least 10 pack years.

Exclusion Criteria:

* Patients who have not achieved acceptable spirometry results at run-in, in accordance with American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria for acceptability and repeatability.
* Patients who have had 2 or more COPD exacerbations that required treatment with antibiotics, systemic steroids (oral or intravenous) or hospitalization in the 12 months prior to Visit 1.
* Patients who have had a respiratory tract infection.
* Patients requiring long-term oxygen therapy (>12 hours a day) on a daily basis.
* Patients with a) any history of asthma, or b) onset of respiratory symptoms prior to age 40 years.
* Patients with allergic rhinitis who use a H1-antagonist or intra-nasal corticosteroids intermittently. Treatment with a stable dose is permitted.
* Patients with concomitant pulmonary disease (e.g., lung fibrosis, sarcoidosis, interstitial lung disorder, pulmonary hypertension) or active pulmonary tuberculosis
* Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy comparison of indacaterol to placebo | 12 weeks
  Efficacy comparison of indacaterol to placebo (once daily treatment) by measuring Trough Forced Expiratory Volume in one second 24 hour postdose after 12 weeks of treatment.

SECONDARY OUTCOMES:
St George's Respiratory Questionnaire for COPD (SGRQ- C) total score comparison between treatments | 12 weeks
  Effects comparison of indacaterol to placebo in terms of the patient-centric measurement St George's Respiratory Questionnaire for COPD (SGRQ- C) total score after 12 weeks of treatment.
Comparison of Forced Expiratory Volume in one second between indacaterol and tiotropium groups | 12 weeks
  Comparison of indacaterol to tiotropium using Trough Forced Expiratory Volume in one second.
St George's Respiratory Questionnaire for COPD total score comparison between treatments | 12 weeks
  Effects comparison of indacaterol to tiotropium in terms of St George's Respiratory Questionnaire for COPD (SGRQ- C) total score after 12 weeks of treatment.
Adverse events and serious adverse events for all treatment groups | week 12
  All adverse events will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals